CLINICAL TRIAL: NCT03426371
Title: With or withoutA140 + mFOLFOX6 Treat 1st Line mCRC in RAS Wide Type, Multicenter, Double-blind, Randomized, Controlled Phase III Trial
Brief Title: Epidermal Growth Factor Receptor (EGFR) Antagonist Chimeric Anti-EGFR Monoclonal Antibody Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KL140-III-01
Record Dates: First submitted 2018-01-24; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: multicenter, double-blind, randomized, controlled phase III trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All eligible subjects will receive KL-140 in combination with mFOLFOX-6 chemotherapy regimen.
  Interventions: Drug: KL-140
- Placebo Comparator (Placebo Comparator): All eligible subjects will receive Placebo in combination with mFOLFOX-6 chemotherapy regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KL-140 — KL-140 will be administered every 7 days at an initial dose of 400 milligram per square meter (mg/m^2) at 5 milligram per minute (mg/min) and 250 mg/m^2 at 10 mg/min for subsequent infusions until progression of disease, withdrawal of consent, or unacceptable toxicity to KL-140.
  Drug: Oxaliplatin Oxaliplatin 85 mg/m^2 infusion over 120 minutes on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Drug: Folinic Acid FA 200 mg/m^2 infusion over 120 minutes on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Drug: 5Fluorouracil 5-FU as a bolus of 400 mg/m^2/day intravenously followed by 2400 mg/m^2/day infusion over 48 hours on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Arms: Experimental
Drug: Placebo — Placebo will be administered every 7 days at an initial dose of 400 milligram per square meter (mg/m^2) at 5 milligram per minute (mg/min) and 250 mg/m^2 at 10 mg/min for subsequent infusions until progression of disease, withdrawal of consent, or unacceptable toxicity Drug: Oxaliplatin Oxaliplatin 85 mg/m^2 infusion over 120 minutes on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Drug: Folinic Acid FA 200 mg/m^2 infusion over 120 minutes on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Drug: 5Fluorouracil 5-FU as a bolus of 400 mg/m^2/day intravenously followed by 2400 mg/m^2/day infusion over 48 hours on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Arms: Placebo Comparator

SUMMARY:
The study is an double blind, randomized, multicenter phase 3 trial. The efficacy analyses are based on 570 Chinese patients with RAS wt mCRC treated with mFOLFOX-6 ± cetuximab. Study treatment continues until disease progression or unacceptable toxicity (ie, not for a fixed number of courses). The primary endpoint of the study is progression-free survival (PFS) time according to RECIST 1.0; key secondary endpoints include overall survival (OS) time, overall response rate (ORR), and safety/tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female subjects， 18-75 years of age
* Medically accepted effective contraception if procreative potential exists
* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* RAS wild-type and BRAF-V600E wild-type status in tumor tissue
* At least one measurable lesion by computer tomography (CT) or magnetic resonance imaging (MRI) according to RECIST
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at trial entry
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at trial entry
* White blood cell count >= 3 × 10x9/L with neutrophils >= 1.5 × 10x9/L, platelet count >=75 × 10x9/L and hemoglobin >= 8 g/dL； Total bilirubin <= 1.5 × upper limit of reference range， Aspartate transaminase (AST) and alanine transaminase (ALT) <= 2.5 × upper limit of reference range or <= 5 × upper reference range in subjects with liver metastasis；Serum creatinine <= 1.5 × upper limit of reference range

Exclusion Criteria:

* Known hypersensitivity or allergic reactions against any of the components of the trial treatments
* Radiotherapy or surgery (excluding prior diagnostic biopsy) in the 28 days before trial treatment
* Known brain metastasis and/or leptomeningeal disease. Subjects with neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasis
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease，except the patient with fistulation or stenting
* Active clinically serious infections (> grade 2 National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0), including active tuberculosis
* Uncontrolled diabetes mellitus, pulmonary fibrosis, acute pulmonary disorder, interstitial pneumonia, or liver failure
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 5 years, or left ventricular ejection fraction below the institutional range of normal on a baseline multiple gated acquisition scan or echocardiogram
* Renal replacement therapy
* Peripheral neuropathy > grade 1
* History of organ allograft, autologous stem cell transplantation, or allogeneic stem cell transplantation
* Previous malignancy other than CRC in the last 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix
* Known and declared history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Known severe coagulation disorders
* Previous chemotherapy for CRC except adjuvant treatment if terminated > 12 months (oxaliplatin-based chemotherapy) or > 6 months (non-oxaliplatin-based chemotherapy) before the start of treatment in this trial
* Previous treatment with anti-EGFR monoclonal antibody therapy
* Other non-permitted concomitant anticancer therapies, chronic systemic immune therapy or hormone therapy
* Granulocyte colony stimulating factor (G-CSF) or granulocyte macrophage colony stimulating factor (GM-CSF) within 3 weeks of trial entry，blood transfusion，or blood components transfusion
* Pregnancy (absence to be confirmed by serum β-human chorionic gonadotropin test) or breastfeeding
* Ongoing alcohol or drug abuse
* Known neurological or psychiatric diseases
* Participation in another clinical trial within the past 4 weeks
* Legal incapacity or limited legal capacity
* Other significant disease that in the investigator's opinion should exclude the subject from the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) Time | Time Frame: Baseline up to 128 weeks
  PFS was defined as the duration (in months) from randomization until the first progressive disease (PD) observation as assessed by the investigators according to Response Evaluation Criteria for Solid Tumors (RECIST) version 1.0, or death due to any cause when death occurred within 90 days of randomization or the last tumor assessment, whichever was later. PD was defined as at least a 20% increase in the sum of longest diameter (LD) of the target lesions, taking as references the smallest sum LD since the treatment started (including baseline), or appearance of one or more new lesions, and/or unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
Overall Survival (OS) Time | Time Frame: Baseline up to 258 weeks
  OS was defined as the time (in months) from randomization to death. For subjects who were still alive at the analysis data cut-off date or who lost to follow-up, survival was censored at the last recorded date that the subject was known to be alive.
Best Overall Response Rate (ORR) | Time Frame: Baseline up to 128 weeks
  The Best ORR was defined as the percentage of subjects having achieved complete response (CR) or partial response (PR) according to RECIST version 1.0 as determined by the IRC. CR: defined as disappearance of all target and all non-target lesions and no new lesions. PR: defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters, no progression of non-target lesions and no new lesions.
  The Best ORR was defined as the percentage of subjects having achieved complete response (CR) or partial response (PR) according to RECIST version 1.0 as determined by the investigators. CR: defined as disappearance of all target and all non-target lesions and no new lesions. PR: defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters, no progression of non-target lesions and no new lesions.
Time to Treatment Failure (TTF) | Time Frame: Baseline up to 128 weeks
  TTF was defined as time from randomization to date of the first occurrence of radiologically confirmed PD. Clinical PD according to the Investigator's assessment , discontinuation of treatment due to progression or adverse event, start of new anticancer therapy, withdrawal of consent, or death within 90 days of last tumor assessment or randomization. Subjects without event were censored on the date of last tumor assessment.
quality of life score | Time Frame: Baseline up to 258 weeks
  Quality of life score is defined of questionnaire EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China